CLINICAL TRIAL: NCT03186118
Title: Pediatric and Young Adult Leukemia Adoptive Therapy (PLAT)-03: A Pilot Feasibility and Safety Study of CD19t T-Antigen Presenting Cells (T-APCs) Following CAR T Cell Immunotherapy for CD19+ Leukemia
Brief Title: Pilot Study of T-APCs Following CAR T Cell Immunotherapy for CD19+ Leukemia
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Colleen Annesley, Medical Director, Seattle Children's Therapeutics, Seattle Children's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PLAT-03
Record Dates: First submitted 2017-06-12; First posted 2017-06-14 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: CD 19+ Acute Leukemia
Keywords: pediatric; young adult; acute lymphoblastic leukemia; CD 19; leukemia; chimeric antigen receptor; T cell
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Intervention Model Description: Subjects are assessed during the parent study for total CD 19 load in bone marrow. Participants meeting eligibility criteria are transitioned into one of 3 arms in PLAT-03.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort A (Experimental): Participants will receive CD19-targeting CAR T cells. Participants who have a total CD19 antigen load in bone marrow of <15% will be assigned to Cohort A, to receive up to 6 T-APC treatments.
  Interventions: Biological: T-cell Antigen Presenting Cells expressing truncated CD19 (T-APC)
- Cohort B (Experimental): Participants will receive CD19-targeting CAR T cells. Participants for whom laboratory testing on Study Day 14 indicates they are at risk for early loss of CAR T cells will be assigned to Cohort B to receive up to 6 T-APC treatments. If laboratory testing prior to planned T-APC treatment indicates loss of CAR-T cells, participants may move to Cohort C.
  Interventions: Biological: T-cell Antigen Presenting Cells expressing truncated CD19 (T-APC)
- Cohort C (Experimental): Participants will receive CD19-targeting CAR T cells. Participants for whom laboratory testing shows loss of CAR T cells within 6 months will be assigned to Cohort C. They will receive another CAR T cell infusion followed by up to 6 T-APC treatments.
  Interventions: Biological: T-cell Antigen Presenting Cells expressing truncated CD19 (T-APC)
- Cohort D (Experimental): Participants will receive CD19-targeting CAR T cells. Participants who do not meet assignment rules for Cohorts A, B, or C will be followed after CAR T cell infusion in Cohort D.
  Interventions: Biological: T-cell Antigen Presenting Cells expressing truncated CD19 (T-APC)

INTERVENTIONS:
Biological: T-cell Antigen Presenting Cells expressing truncated CD19 (T-APC) — Autologous CD4 and CD8 T cells transduced to express a truncated CD19 (CD19t) Transgene
  Other Names: CD19+ Chimeric Antigen Receptor T-cells (CAR-T cells)

SUMMARY:
Patients with relapsed or refractory CD 19+ leukemia who have achieved remission after CD19 CAR-T cell treatment sometimes relapse because the CD 19 CAR-T cells decrease in number over time. Study PLAT-03 will test whether administering T cell antigen presenting cells (T-APCs) at intervals following treatment with CAR-T cells improves CD 19 CAR-T cell persistence and reduces the incidence of leukemia relapse.

DETAILED DESCRIPTION:
This pilot study seeks to examine the feasibility and safety of administering T cell antigen presenting cells (T-APCs) designed to reactivate and numerically expand CD19-specific CAR T cells. The underlying hypothesis to be examined is that after remission is achieved with CAR T cell treatment, the duration, magnitude, and activation state of persisting memory CAR T cells impact on the potential for durable leukemia eradication. This is of particular relevance in two groups of patients we have identified: those who are predicted to lose persistence of their CAR T cells before Day 63, and those who have definitively lost persistence of CAR T cells prior to 6 months. By providing these patients with episodic exposure to T-APCs capable of activating CD19-specific CAR T cells for proliferation and redistribution to tissue beds where tumor cells of ALL seed, ideally over several months following remission induction, it is posited that the incidence of disease relapse will be diminished.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of recurrent or refractory CD19+ leukemia
* Adequate performance status
* Able to tolerate apheresis, including placement of temporary apheresis line if required
* Adequate renal, liver, cardiac, and respiratory function
* Adequate absolute lymphocyte count
* HIV negative; Hepatitis B and C negative within 3 months prior to enrollment.

Exclusion Criteria:

* Evidence of active clinically significant CNS dysfunction
* Evidence of active malignancy other than CD19+ malignancy
* Evidence of active GVHD, or on immunosuppressive GVHD therapy within 4 weeks prior to enrollment

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-08-04 (Actual); Primary Completion 2021-09-13 (Actual); Study Completion 2033-07 (Estimated)

PRIMARY OUTCOMES:
The adverse events associated with one or multiple CD19t T-APC product infusions will be assessed. | up to 6 months
  Type, frequency, severity, and duration of adverse events will be summarized
Determine the feasibility of deriving and administering a CD19t T-APC product | 28 days
  Proportion of products successfully manufactured and infused

SECONDARY OUTCOMES:
Quantification of changes in the number of CAR T cells in peripheral blood before and after receiving CD19t T-APCs | 6 months
  Multiparameter Flow Cytometry (MPF) from peripheral blood as a measure of magnitude and presence of CAR T cells before and after a dose of T-APCs
Duration of B cell aplasia in CD19t T-APC treated patients | up to 5 years
  MPF from peripheral blood as a measure of B cell aplasia

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Annesley, MD, Study Chair — Seattle Children's Hospital
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No
will not be shared

REFERENCES:
- [Derived] Annesley C, Seidel K, Wu Q, Summers C, Wayne AS, Pulsipher MA, Agrawal AK, Brown CT, Mgebroff S, Lindgren C, Rawlings-Rhea S, Huang W, Wilson AL, Jensen MC, Park JR, Gardner RA. Outcomes of PLAT-02 and PLAT-03: evaluating CD19 CAR T-cell therapy and CD19-expressing T-APC support in pediatric B-ALL. Blood. 2025 Aug 14;146(7):789-801. doi: 10.1182/blood.2025028359. PMID 40233328